CLINICAL TRIAL: NCT05439863
Title: Transcatheter Aortic Valve Replacement for Severe Aortic Valve Disease: Multi-center, Real-word Registry
Brief Title: TAVR for Aortic Valve Disease
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Junjie Zhang, Vice chief, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: NanjingValve Registry
Record Dates: First submitted 2022-05-27; First posted 2022-06-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVR in aortic valve disease
  Interventions: Device: transcatheter heart valve

INTERVENTIONS:
Device: transcatheter heart valve — patients with severe aortic valve disease underwent transcatheter heart valve

SUMMARY:
Transcatheter aortic valve replacement (TAVR) has became an important treatment of severe aortic stenosis (AS). Several randomized clinical trials showed that TAVR was non-inferior or superior to surgical aortic valve replacement (SAVR). However, many different issues have emerged: TAVR in younger patients? valve leaflet thrombosis? transcatheter valve durability? coronary reaccess after TAVR? TAVR in bicuspid aortic valve? TAVR in aortic regurgitation? etc. Hence, a prospective, multicenter database is created to provide the real-word data for these questions.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of severe aortic stenosis or aortic regurgitation
2. Patients undergo transcatheter aortic valve replacement

Exclusion Criteria:

patients refuse the clinical follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing transcatheter aortic valve replacement due to severe aortic valve stenosis or regurgitation were eligible into this registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2032-12-30 (Estimated); Study Completion 2037-12-30 (Estimated)

PRIMARY OUTCOMES:
all-cause death during follow-up | 5 years
  all-cause death during 5-year follow-up

SECONDARY OUTCOMES:
cardiac death during follow-up | 5 years
  Cardiac death during 5-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No